CLINICAL TRIAL: NCT05739656
Title: A PROSPECTIVE, MULTICENTER, POST-MARKET OBSERVATIONAL STUDY TO EVALUATE ROTATIONAL STABILITY AND FUNCTIONAL VISUAL ACUITY OF THE ENVISTA ONE-PIECE HYDROPHOBIC ACRYLIC TORIC IOL MX60ET FOLLOWING CATARACT SURGERY PROTOCOL.
Brief Title: Evaluation of Visual Acuity of the Envista One-piece Acrylic Toric IOL MX60ET
Status: Completed | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 897
Record Dates: First submitted 2023-01-17; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: CATARACT SURGERY — Approximately up to 100 subjects (100 eyes) will be successfully implanted with an enVista Toric IOL (Model MX60ET) in one or both eyes.
  Other Names: The enVista One-Piece Hydrophobic Acrylic Toric IOL

SUMMARY:
The primary objective of this study is to evaluate rotational stability and functional improvements in visual acuity of the enVista monofocal Toric IOL (MX60ET) following cataract surgery.

DETAILED DESCRIPTION:
This is a prospective, multicenter, post-market observational study at approximately 5 sites in the United States. All clinical sites will have Institutional Review Board (IRB) approval prior to recruiting potential subjects. All subjects who meet eligibility criteria will be consecutively offered enrollment into the trial. Approximately up to 100 subjects (100 eyes) will be successfully implanted with an enVista Toric IOL (Model MX60ET) in one or both eyes at up to 5 clinical sites in the United States. For subjects with pre-existing cataracts in both eyes requiring removal and IOL implantation, the eye with the worse BCDVA at the preoperative visit will be designated the study eye. If BCDVA is the same for both eyes, the right eye will be designated the study eye. Postoperatively, all subjects will undergo ophthalmic examinations at regular intervals per the study visit schedule through Form 4 (120-180 days postoperative).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to read, understand, and provide written informed consent on the Institutional Review Board (IRB)-approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.
* Subjects must be able and willing to comply with all treatment and follow-up/study procedures.
* Subjects must be 18 years of age or older on the date the ICF is signed.
* Subjects must have best-corrected distance visual acuity (BCDVA) equal to or worse than 20/40 in the study eye, with or without glare source, due to a clinically significant cataract (either cortical, nuclear, subcapsular, or a combination) that is considered amenable to treatment with standard phacoemulsification cataract extraction.
* Subjects must require a spherical equivalent lens power from 17.0 D to 24.0 D in the study eye.
* Subjects must have a BCDVA projected to be better than 20/30 after toric IOL implantation in the study eye (as determined by the medical judgment of the Investigator or measured by potential VA testing if necessary).
* Subjects must have a preoperative corneal astigmatism between 0.77 D and 4.53 D in the study eye.
* Subject must have a dilated preoperative pupil size greater than or equal to 5.0 mm in the study eye.
* Contact lens wearers need to demonstrate a stable refraction (within

  ±0.50 D) in the study eye, as determined by manifest refraction spherical equivalent (MRSE) on two consecutive examination dates. Stability of the refraction is determined under the following conditions:

  - Lenses are not worn for at least 2 weeks (rigid or toric contact lenses) or 3 days (soft contact lenses) prior to the first refraction used to establish stability and through the day of surgery.
* The two refractions are performed at least 7 days apart.

Exclusion Criteria:

This study will exclude subjects who meet none of the following exclusion criteria:

* Subjects with any anterior segment pathology in the study eye likely to increase the risk of complications from phacoemulsification cataract surgery (eg, chronic uveitis, iritis, iridocyclitis, rubeosis iridis, clinically significant corneal dystrophy, clinically significant Fuchs' dystrophy, clinically significant anterior membrane dystrophy, etc).
* Subjects with associated ocular conditions which could affect the stability of the IOL (eg, traumatic zonulolysis, zonular dialysis, evident zonular weakness or dehiscence, etc) in the study eye.
* Subjects with clinically significant irregular corneal astigmatism in the study eye, as determined by the medical judgment of the Investigator.
* Subjects with clinically significant corneal pathology potentially affecting topography of either eye.
* Subjects with any ocular condition (eg, amblyopia) that could prevent the possibility of a visual outcome better than 20/30 in the study eye.
* Subjects with an anterior chamber depth < 2.0 mm as measured by the IOL master/LENSTAR in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately up to 100 subjects (100 eyes) will be successfully implanted with an enVista Toric IOL (Model MX60ET) in at least one eye. For subjects with pre-existing cataracts in both eyes requiring removal and IOL implantation, the eye with the worse BCDVA at the preoperative visit will be designated the study eye. If BCDVA is the same for both eyes, the right eye will be designated the study eye. Only the study eye data will be collected, and binocular visual acuities will not captured. Postoperatively, all subjects will undergo ophthalmic examinations at regular intervals per the study visit schedule through Form 4 (120-180 days postoperative).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | The duration of the study, including the time to recruit all subjects, will be up to 12 months. Eligible subjects who are enrolled in the study will be seen for up to 6 months after implantation.
  The proportion of subjects with absolute lens axis rotation from surgical placement of less than or equal to 20 degrees. Tertiary/Supportive/Other effectiveness outcomes will include the following.
  * Uncorrected and distance-corrected visual acuities at 66 cm and at 4 m
  * Manifest refraction
  * Subjective questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Jeffrey Whitman, MD, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holladay JT, Haller M. Light Adjustable Lens Results of Spherical Equivalent and Astigmatism Correction from the FDA Post-Approval Study. J Cataract Refract Surg. 2026 Feb 10. doi: 10.1097/j.jcrs.0000000000001906. Online ahead of print. PMID 41664266